CLINICAL TRIAL: NCT06116695
Title: Tomographic Evaluation of Apexogenesis With Human Treated Dentin Matrix in Young Permanent Molars
Brief Title: Tomographic Evaluation of Pulpotomy in Young Permanent Teeth Using Human-treated Dentin Matrix
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, nora mostafa mohammed abo shanady, Assistant lecturer at pediatric dentistry oral health and preventive dentistry department, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-21-1
Record Dates: First submitted 2023-10-27; First posted 2023-11-03 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Pulpotomy of Young Permanent Molars
MeSH Terms: interventions — TheraCal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- human-treated dentin matrix (Experimental): drug: Human-treated dentin matrix young permanent molars treated with human-treated dentin matrix
  Interventions: Drug: human treated dentin matrix
- mineral tri oxide aggregate (Placebo Comparator): Drug: Mineral Trioxide Aggregate young permanent molars treated with Mineral Trioxide Aggregate mineral trioxide aggregate was used as control
  Interventions: Drug: Mineral Tri-Oxide Aggregate

INTERVENTIONS:
Drug: human treated dentin matrix — human treated dentin matrix is compared with mineral trioxide aggregate in apexogenesis
  Other Names: human partially demineralized treated dentin matrix
  Arms: human-treated dentin matrix
Drug: Mineral Tri-Oxide Aggregate — mineral trioxide aggregate was used as control
  Arms: mineral tri oxide aggregate

SUMMARY:
Assess tomographic outcomes of pulpotomy in young permanent molars using human-treated dentin matrix versus MTA.

DETAILED DESCRIPTION:
The study was conducted as a split-mouth randomized clinical trial, approved by research ethics committee, Faculty of Dentistry, Tanta University, and carried out at Pediatric Dentistry Department, Faculty of Dentistry, Tanta University. The material preparation was conducted at Pharmaceutical Technology Department, Faculty of Pharmacy, Tanta University. 20 children of both sexes aged from 6 to 8 years old were selected with bilateral deeply carious young permanent mandibular first molars that are indicated for pulpotomy procedure.The selected deeply carious molars were randomly divided into two groups as follows:

Group I (Study group): 20 molars were treated with hTDM. Group II:

(Control group): 20 molars were treated with White MTA. The participating cases were evaluated clinically 3, 6, 12 and 18 months. Digital periapical radiographs was taken at 6 month follow-up period to ensure the state of the treated teeth or if there was necessary condition.

Tomographic evaluation was performed immediate postoperatively and at 18 months.

ELIGIBILITY:
Inclusion Criteria:.

1. Bilateral immature permanent mandibular first molars with deep carious lesions.
2. Positive response to pulp testing.
3. Normal radiographic appearance.
4. Healthy children without any systemic disease that interferes with pulp healing.
5. Patient and parent cooperation.

Exclusion Criteria:

1. Clinical signs and symptoms of irreversible pulpitis as spontaneous throbbing pain, tenderness to percussion, abnormal tooth mobility, swelling, or sinus tract.
2. Presence of periapical lesion, external or internal root resorption.
3. Carious furcation involvement.
4. Dystrophic calcification of the pulp.
5. Non restorable tooth.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-06-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
clinical outcomes | 18 months
  Absence of pain related to the treated teeth, including pain or sensitivity to percussion/palpation, No evidence of swelling or presence of a sinus tract, Absence of mobility affecting the treated teeth
Tomographic outcomes | 18 months
  Continuous increase in root length and decrease in the apical diameter, Absence of radicular, interradicular and periradicular rarefaction, No loss of the lamina dura.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Tanta University, Tanta, El Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Li R, Guo W, Yang B, Guo L, Sheng L, Chen G, Li Y, Zou Q, Xie D, An X, Chen Y, Tian W. Human treated dentin matrix as a natural scaffold for complete human dentin tissue regeneration. Biomaterials. 2011 Jul;32(20):4525-38. doi: 10.1016/j.biomaterials.2011.03.008. Epub 2011 Mar 31. PMID 21458067
- [Result] Tabatabaei FS, Tatari S, Samadi R, Torshabi M. Surface characterization and biological properties of regular dentin, demineralized dentin, and deproteinized dentin. J Mater Sci Mater Med. 2016 Nov;27(11):164. doi: 10.1007/s10856-016-5780-8. Epub 2016 Sep 21. PMID 27655430
- [Result] Widbiller M, Eidt A, Wolflick M, Lindner SR, Schweikl H, Hiller KA, Buchalla W, Galler KM. Interactive effects of LPS and dentine matrix proteins on human dental pulp stem cells. Int Endod J. 2018 Aug;51(8):877-888. doi: 10.1111/iej.12897. Epub 2018 Feb 17. PMID 29377169
- [Result] Chen J, Cui C, Qiao X, Yang B, Yu M, Guo W, Tian W. Treated dentin matrix paste as a novel pulp capping agent for dentin regeneration. J Tissue Eng Regen Med. 2017 Dec;11(12):3428-3436. doi: 10.1002/term.2256. Epub 2017 Feb 15. PMID 28198096
- [Derived] Shanady NMA, Abo Hamila NA, El Maghraby GM, Ghouraba RF. Tomographic evaluation of apexogenesis with human treated dentin matrix in young permanent molars: a split-mouth randomized controlled clinical trial. BMC Oral Health. 2025 May 7;25(1):692. doi: 10.1186/s12903-025-05997-1. PMID 40335983